CLINICAL TRIAL: NCT07265999
Title: Severity Factors of Dermatomyositis in the Caribbean Population - DM-ANTILLES
Acronym: DM-ANTILLES
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH3_2020/11
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Dermatomyositis
Keywords: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Additional blood samples required for research, including HLA typing and serum interferon assays, will consist of up to three 3.5 mL dry tubes and one 5 mL EDTA tube (total 15.5 mL).
  HLA typing samples (1 × 5 mL EDTA tube) will be transported internally to the CHU Guadeloupe Immuno-Hematology Laboratory for processing.
  Serum interferon samples (3 × 3.5 mL tubes) will be sent to the CHU Guadeloupe Biobank (CRB), centrifuged, aliquoted into cryotubes, and stored at -80 °C until batch shipment to the processing site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with dermatomyositis: All patient with dermatomyositis

SUMMARY:
Dermatomyositis is a rare chronic autoimmune and inflammatory disease that affects the skin and striated muscles. Its prognosis is linked to visceral involvement (lungs, heart, and oropharyngeal region) and to the possible presence of associated cancer. The implementation of the research will allow identification of incident cases of dermatomyositis in Guadeloupe and the characterization of the disease in the overseas population, in the absence of data in the literature.

DETAILED DESCRIPTION:
In the French West Indies, this condition is associated with high short- and medium-term morbidity and mortality. Diagnostic delays and patient care pathways may help explain this. However, a particularly severe phenotype of the disease in Antillean patients may also play a role, as observed in other autoimmune and inflammatory diseases we have described in overseas populations (e.g., systemic sclerosis, sarcoidosis).

Identifying factors associated with the severity of dermatomyositis at the time of diagnosis would allow for the early implementation of a tailored management strategy to improve the disease prognosis in the target population.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of dermatomyositis according to the 2003 ENMC criteria
* Patient with parents or grandparents originating from the Caribbean arc
* Patient aged 16 years or older
* Patient residing in Guadeloupe
* Patient (or legal representative) who has received information about the study and has signed the informed consent form
* Patient affiliated with a social security scheme

Exclusion Criteria:

* Patient who started treatment with intravenous immunoglobulins, corticosteroids, or immunosuppressants within the month prior to the diagnosis of dermatomyositis
* Patient under legal protection (guardianship or trusteeship) or deprived of liberty

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients (>16 years old) diagnosed with dermatomyositis, including both classic dermatomyositis and clinically amyopathic dermatomyositis, regardless of sex or ethnicity. Eligible patients are those who have received a new diagnosis and can be followed for at least two years.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2029-07-16 (Estimated); Study Completion 2029-07-16 (Estimated)

PRIMARY OUTCOMES:
severity of dermatomyositis at diagnosis | Assessed at baseline (diagnosis).
  The primary outcome measure is the severity of dermatomyositis at diagnosis, defined by the presence of one or more of the following criteria:
  Muscle involvement resulting in functional disability; Associated visceral involvement, including the heart, lungs, or oropharyngeal region; Associated cancer, either previously diagnosed within the past three years or diagnosed concurrently with dermatomyositis.

SECONDARY OUTCOMES:
Mortality | Assessed over 2 years from the date of dermatomyositis diagnosis
  Number of participants who die from any cause during the follow-up period.
  Units: Count of participants
Relapse Occurrence | Assessed over 2 years from the date of dermatomyositis diagnosis
  Number of participants experiencing relapse(s) during treatment tapering or after treatment discontinuation.
  Units: Count of participants
Cancer Occurrence | Assessed over 2 years from the date of dermatomyositis diagnosis
  Number of participants diagnosed with any cancer during the follow-up period.
  Units: Count of participants

CONTACTS AND LOCATIONS:
Overall Officials: nadège cordel, MD PhD, Principal Investigator — CHU de la Guadeloupe
Locations (1):
- CHU de la Guadeloupe, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No